CLINICAL TRIAL: NCT06259799
Title: Efficacy of a Smart Water Bottle Intervention to Increase Fluid Consumption in College Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kennesaw State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MZ
Record Dates: First submitted 2024-02-07; First posted 2024-02-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Dehydration
Keywords: underhydration; copeptin; urine; water
MeSH Terms: conditions — Dehydration; Diabetes Insipidus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart Water Bottle (Experimental): Participants in the intervention group will be prompted by the water bottle to drink (bottle will light up red) whenever they are behind on fluid intake recommendations for the day. The bottle will be linked to a smart phone application that participants will be instructed to download on their personal mobile device, but they will log into this device using a researcher provided username and password. The bottle will encourage male participants to consume 2.5 L and for female participants to consume 2.0 L of fluid. Participants will be asked to use this bottle to consume all water and enter any additional sources of fluid using the mobile application. The intervention group will also be asked to record their daily perceived thirst, first morning urine color, and body mass as a means of self-monitoring daily changes in hydration status, using a provided paper log.
  Interventions: Behavioral: Smart Water Bottle
- Control (No Intervention): The control group will be asked to go about daily activities as normal. They will not receive the water bottle and will not be asked to track daily measures of thirst, morning urine color, or body mass.

INTERVENTIONS:
Behavioral: Smart Water Bottle — Participants in the intervention group will receive a bottle which measures participant fluid consumption. The bottle will be set to recommend 2.5L for male participants and 2.0L for female participants, consistent with fluid intake recommendations from the European Food Safety Authority for each sex. Participants will be prompted by the bottle (bottle will light up) when they are behind on fluid intake recommendations. Participants will use a validated urine color chart, 9 point Likert scale for thirst, and measure nude body mass on their own each morning. Participants will be informed that higher values for nude body mass and thirst, and lower values for nude body mass each morning may indicate they are less hydrated day-to-day.
  Arms: Smart Water Bottle

SUMMARY:
Approximately 60% of males and 40% of females do not meet current fluid intake recommendations, which is associated with adverse health consequences such as obesity, diabetes, and chronic kidney disease. Newer technologies have been designed to promote fluid intake. "Smart Water Bottles" use mHealth technology to capture fluid intake behaviors automatically and provide cues to encourage fluid consumption. Studies using Smart Water Bottles have helped some individuals increase fluid intake to help reduce kidney stone formation. However, limited research has assessed the efficacy of this technology on improving fluid intake in college students. College is a time with the potential to form healthy habits that carry into adulthood. Previous work has also identified daily changes in morning urine color, thirst perception, and body mass, as simple, inexpensive indicators of daily fluctuations in water balance. Tracking changes in these metrics has the potential to provide participants with evidence of adequate or inadequate fluid consumption. Thus, the combination of prompting from a smart water bottle, as well as daily self-monitoring changes in hydration status, may encourage college students to increase daily fluid consumption.

ELIGIBILITY:
Inclusion Criteria:

* Participants must report currently drinking less than the European Food Safety Authority Recommendations for fluid, as determined by an online pre-screening survey (<2.5 L per day for males; <2.0 L per day for females).
* Has access to a cell phone which can download the app associated with the Smart Water Bottle.

Exclusion Criteria:

* Currently trying to gain or lose weight
* Have had surgery of the digestive tract
* Currently taking diuretics (e.g., Thiazide, Loop diuretics or potassium-sparing diuretics)
* Currently taking centrally-acting medications (e.g., anesthetics, anticonvulsants, central nervous system stimulants/amphetamines, muscle relaxants)
* Report currently consuming at least the European Food Safety Authority Recommendations for fluid, as determined by an online pre-screening survey (>= 2.5 L per day for males, >=2.0 L per day for females).
* Currently pregnant (females)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Total Fluid Intake | Pre and Post 2-week intervention
  Total Fluid Intake will be reported by participants for 3 days before and after the intervention using a validated fluid log. The average of 3-days of fluid recording will be used.
Changes in 24h urine osmolality | Pre and Post 2-week intervention
  Urinary osmolality reflects the concentration of urine, with higher values indicative of worse hydration. Urine osmolality will be collected for 3 days at the start and end of the study, with the average of each 3 day period used for analyses.
Changes in 24h urine volume | Pre and Post 2-week intervention
  Higher urine volume tends to correspond with greater fluid intake.

SECONDARY OUTCOMES:
Change in urine color measured by validated urine color chart | Pre and Post 2-week intervention
  A validated urine color will be used to rate urine samples. Higher values correspond with worse hydration.
Changes in calorie intake from dietary log. | Pre and Post 2-week intervention
  The ASA-24 is an electronic diet log participants will use to record their diet at the start and end of the study.
Change in copeptin | Pre and Post 2-week intervention
  Copeptin is a surrogate marker for vasopressin, a major fluid regulatory hormone which increases fluid conservation at the kidneys.
Change in urine specific gravity | Pre and Post 2-week intervention
  Measures the density of the urine.
Change in body water distribution | Pre and Post 2-week intervention
  Intracellular and extracellular water content measured via BIA.
Change in Aldosterone | Pre and Post 2-week intervention
  Fluid regulatory hormone involved in plasma volume regulation.
Hydration KAB Scales | Pre and Post 2-week intervention.
  Brief questionnaire assessing hydration knowledge, attitudes, and beliefs about hydration and fluid intake behaviors.
Change in body fat percentage | Pre and Post 2-week intervention
  Assessed via dual-energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

IPD SHARING:
Plan to Share IPD: No